CLINICAL TRIAL: NCT04045509
Title: Investigation in Variability and Repeatability of Corneal Sensation in a Normal Population
Brief Title: Investigation in Corneal Sensation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Daniela Nosch (Other)
Responsible Party: Sponsor-Investigator, Daniela Nosch, Clinical Professor, University of Applied Sciences and Arts Northwestern Switzerland
Organization: University of Applied Sciences and Arts Northwestern Switzerland (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2019-01252
Record Dates: First submitted 2019-07-30; First posted 2019-08-05 (Actual); Last update posted 2019-12-06 (Actual); Status verified 2019-12

CONDITIONS: Cornea; Sense Loss
Keywords: corneal sensation; subbasal nerve plexus
MeSH Terms: conditions — Corneal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 'young age' (Other): Group 'young age': 18 - 30 years of age; healthy eyes
  Interventions: Device: Liquid Jet Esthesiometer Prototype; Device: Tactile Esthesiometer Prototype; Device: Cochet Bonnet esthesiometer
- Group 'advanced age' (Other): Group 'advanced age': 50 - 70 years of age; healthy eyes
  Interventions: Device: Liquid Jet Esthesiometer Prototype; Device: Tactile Esthesiometer Prototype; Device: Cochet Bonnet esthesiometer

INTERVENTIONS:
Device: Liquid Jet Esthesiometer Prototype — Balanced salt solution with a pH value similar to the tear film uesd as a liquid jet stimulus for corneal sensation threshold measurement
Device: Tactile Esthesiometer Prototype — A round plastic nozzle (1.8mm diameter) used as a stimulus for corneal sensation threshold measurement
Device: Cochet Bonnet esthesiometer — A nylon thread (0.12mm diameter) used as a stimulus for corneal sensation threshold measurement

SUMMARY:
The aim is to find out more about how corneal sensory fibres react to different types of stimuli (liquid / tactile / nylon thread) and how this can be consciously perceived by the individual. Is it possible to generate a stimulus that delivers a repeatable and reliable response within a useful stimulus force range which allows an interpretation / evaluation of normal / expected activity of superficial nerve fibres in the cornea? The study group will be divided into two age groups, as sensitivity changes are thought to occur in dependence of age. In vivo confocal microscopy has shown that the density of corneal nerve fibres in the sub-basal nerve plexus decreases with age, which consequently would suggest that sensitivity should also decrease. A very interesting research question is to find out, if such sensitivity differences can be detected with the nature of the stimuli applied in this study.

DETAILED DESCRIPTION:
The aim of this study is to gain more physiological knowledge about ocular surface sensation (corneal sensitivity), with application of three different concepts employing different types of stimuli for triggering a response from the pain sensitive nerve endings in the superficial cornea: 1) liquid jet (consisting of isotonic saline solution; prototype), 2) tactile stimulus (round plastic nozzle, prototype) 3) commercially available Cochet Bonnet esthesiometer (nylon thread). Measurements will be carried out on healthy eyes of subjects in two different age groups.

Current knowledge about human corneal sensitivity is limited, as applied methods for ocular surface sensation measurement are limited with regards to reproducibility / accuracy.

Corneal sensitivity represents a neurological response from the free nerve endings within the epithelium. They are sensitive to mechanical, electrical, chemical or thermal stimuli and hence have a protective function for the cornea. Corneal nerves play an important role in cell growth and proliferation of epithelial cells, wound healing and repair. In experimental studies, corneal denervation has been reported to result in epithelial changes: increased permeability, decreased proliferation, changed appearance and delayed wound healing. Therefore, intact corneal innervation is required to maintain the integrity of a normal corneal epithelium. Corneal sensory nerves are believed to play an important role in maintaining the resting tear flow, as their afferent impulses from the ocular surface lead to a reflex response, best described by the lacrimal functional unit: an integrated system comprising the ocular surface tissues (cornea, corneal limbus, conjunctiva, conjunctival blood vessels, and eyelids), the tear secreting components (main and accessory lacrimal glands, meibomian glands, conjunctival goblet, and epithelial cells), and the sensory and motor nerves that connect them.

Current knowledge about ocular surface sensitivity is insufficient, as currently available measurement possibilities lack repeatability and accuracy. Before a new instrument can be developed, more research is required, in order to find a suitable concept for precise sensitivity measurement. For this purpose, two new different concepts with different / new stimulus types will be applied repeatably on healthy eyes in this study. The aim is to find out more about how corneal sensory fibres react to different types of stimuli (liquid / tactile / nylon thread) and how this can be consciously perceived by the individual. Is it possible to generate a stimulus that delivers a repeatable and reliable response within a useful stimulus force range which allows an interpretation / evaluation of normal / expected activity of superficial nerve fibres in the cornea? The study group will be divided into two age groups, as sensitivity changes are thought to occur in dependence of age. In vivo confocal microscopy has shown that the density of corneal nerve fibres in the sub-basal nerve plexus decreases with age, which consequently would suggest that sensitivity should also decrease. A very interesting research question is to find out, if such sensitivity differences can be detected with the nature of the stimuli applied in this study.

ELIGIBILITY:
Inclusion Criteria:

* Group 'young age': 18 - 30 years of age; healthy eyes with Ocular Surface Disease Index Score </= 13
* Group 'advanced age': 50 - 70 years of age; healthy eyes with Ocular Surface Disease Index Score </= 13

Exclusion Criteria:

* Systemic disease that may affect ocular health, such as diabetes
* Injury and history of operations on the anterior segment of the eye
* regular application of systemic or ocular medication known to affect the tear film, specifically on the day of measurement
* rigid gas permeable contact lens wear
* soft contact lens wear less than 48 hours before study visit

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 90 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Repeatability of mechanical corneal sensation thresholds with the Cochet Bonnet esthesiometer | two weeks
  Evaluation of repeatability of mechanical corneal sensation thresholds for the measurement with the Cochet Bonnet instrument (in mN): the corneal sensation thresholds will be obtained with the double staircase method (with forced choice) and the stimulus represents a nylon thread, whereby its force is proportional to the length of the nylon thread applied to the corneal surface.
Repeatability of mechanical corneal sensation thresholds with the liquid jet protoype esthesiometer | two weeks
  Evaluation of repeatability of mechanical corneal sensation thresholds for the measurement with the liquid jet esthesiometer prototype instrument (in mbar): the corneal sensation thresholds will be obtained with the double staircase method (with forced choice) and the stimulus represents a liquid jet (consisting of isotonic saline solution).
Repeatability of mechanical corneal sensation thresholds with the tactile prototype esthesiometer | two weeks
  Evaluation of variability / repeatability of mechanical corneal sensation thresholds for the measurement with the tactile esthesiometer prototype instrument (in mN): the corneal sensation thresholds will be obtained with the double staircase method (with forced choice) and the stimulus represents a small, round plastic ball.

SECONDARY OUTCOMES:
Correlation between corneal sensation thresholds with the Cochet Bonnet esthesiometer | one day
  Correlation between corneal sensitivity thresholds (in mN) obtained with the Cochet Bonnet esthesiometer
Correlation between corneal sensation thresholds with the liquid jet prototype esthesiometer | one day
  Correlation between corneal sensitivity thresholds (in mbar) obtained with the liquid jet prototype esthesiometer
Correlation between corneal sensation thresholds with the tactile prototype esthesiometer | one day
  Correlation between corneal sensitivity thresholds (in mN) obtained with the tactile prototype esthesiometer
Correlation between corneal sensitivity thresholds, obtained with the Cochet Bonnet esthesiometer, and general pain perception | within two weeks
  Correlation between corneal sensitivity thresholds obtained with the Cochet Bonnet esthesiometer and general pain perception, obtained with three different stimulus types, for each of the two different age groups recruited.
Correlation between corneal sensitivity thresholds, obtained with the liquid jet prototype esthesiometer, and general pain perception | within two weeks
  Correlation between corneal sensitivity thresholds, obtained with the liquid jet prototype esthesiometer, and general pain perception
Correlation between corneal sensitivity thresholds, obtained with the tactile prototype esthesiometer, and general pain perception | within two weeks
  Correlation between corneal sensitivity thresholds, obtained with the tactile prototype esthesiometer, and general pain perception
Comparison of corneal sensation thresholds, obtained with the Cochet Bonnet esthesiometer, between the two different age groups in the study population | within two weeks
  Comparison of corneal sensation thresholds obtained with the Cochet Bonnet esthesiometer between the two different age groups in the study population
Comparison of corneal sensation thresholds, obtained with the liquid jet prototype esthesiometer, between the two different age groups in the study population | within two weeks
  Comparison of corneal sensation thresholds, obtained with the liquid jet prototype esthesiometer, between the two different age groups in the study population
Comparison of corneal sensation thresholds, obtained with the tactile prototype esthesiometer, between the two different age groups in the study population | within two weeks
  Comparison of corneal sensation thresholds, obtained with the tactile prototype esthesiometer, between the two different age groups in the study population

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Optometry, FHNW, Olten, Canton of Solothurn, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Nosch DS, Kaser E, Bracher T, Joos RE. Clinical application of the Swiss Liquid Jet Aesthesiometer for corneal sensitivity measurement. Clin Exp Optom. 2024 Jan;107(1):14-22. doi: 10.1080/08164622.2023.2191782. Epub 2023 Apr 5. PMID 37019837